CLINICAL TRIAL: NCT00947986
Title: Effect of Baby Shampoo Nasal Irrigation on Mucociliary Clearance Time in Patients After Sinus Surgery
Brief Title: Mucociliary Clearance Time in Chronic Rhinosinusitis (CRS) Patients After Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Mark Jeffry Amsbaugh, MSII, The University of Texas Medical School at Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-09-0305
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2010-03-22 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Johnson's Baby Shampoo (Experimental): 1% diluted solution
  Interventions: Other: 1% Johnson's Baby Shampoo

INTERVENTIONS:
Other: 1% Johnson's Baby Shampoo — nasal irrigation 2x a day for 4 weeks

SUMMARY:
The investigators are looking at the effects of baby shampoo nasal irrigation on the movement of mucous in the nose in patients who have undergone sinus surgery for chronic sinus problems.

ELIGIBILITY:
Inclusion Criteria:

* CRS
* s/p sinus surgery

Exclusion Criteria:

* nasal polyps

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in mucociliary clearance time (MCT) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UT Department of Otolaryngology Clinic, Houston, Texas, United States